CLINICAL TRIAL: NCT01439620
Title: Pilot Study to Evaluate Optical Frequency Domain Imaging (OFDI) for Biliary Stricture Imaging
Brief Title: Optical Frequency Domain Imaging (OFDI) for Biliary Stricture Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-P-000794
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Biliary Stricture
Keywords: Biliary Stricture; OCT; Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OFDI imaging (Experimental): Subject will swallow an OFDI capsule and images will be obtained using MGH Optical Frequency Domain Imaging (OFDI) imaging system.
  Interventions: Device: MGH Optical Frequency Domain Imaging (OFDI)

INTERVENTIONS:
Device: MGH Optical Frequency Domain Imaging (OFDI) — Imaging of biliary tract with OFDI system using MGH Optical Frequency Domain Imaging (OFDI) System

SUMMARY:
The goal of this study is to evaluate the potential of comprehensive biliary Optical Frequency Domain Imaging (OFDI) for assessing common bile duct or common hepatic duct strictures, determining cholangiocarcinoma margins, and evaluating primary sclerosing cholangitis (PSC).

DETAILED DESCRIPTION:
The study will be conducted in approximately 20 patients with known or suspected common bile duct or common hepatic duct stricture scheduled for endoscopic retrograde cholangiopancreatography (ERCP) with duodenoscope-assisted cholangiopancreatoscopy (DACP) and biopsy.

Following initial fluoroscopic evaluation, the study experimental procedure will begin. The catheter will be passed through the auxiliary channel of the duodenoscope, across the papilla and into the common bile duct. The extra-biliary portion of the catheter will be visible by the duodenoscope at all times. The intrabiliary portion of the catheter will be visible by fluoroscopy, and will be positioned across the biliary stricture. Rotational cross-sectional images of the bile duct will be obtained using the OFDI imaging catheter while pulling back the internal optical components over a pre-determined length. OFDI imaging will be conducted approximately from 1 cm distal to 1 cm and proximal to the stricture margins identified by fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 and up to 75 years old
* Patients able to give informed consent
* Patients with bile duct measuring ≥4 mm in diameter
* Patients with established biliary enteric access - specifically, a previously performed biliary sphincterotomy, or a biliary sphincterotomy performed during the current ERCP for indications other than participation in the study
* Women of childbearing potential must have a negative urine pregnancy test obtained prior to the procedure

Exclusion Criteria:

* Patients with pancreatitis
* Pregnant women
* Patients on oral anticoagulant (warfarin) therapy
* Patients with known history of hemostatic disorder
* Patients found to have a biliary fistula on diagnostic ERCP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2009-07-20 (Actual); Study Completion 2010-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD PhD, Principal Investigator — Massachusetts General Hospital; David Forcione, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OFDI Imaging
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Seven subject were enrolled and completed this study
Arm/Group | OFDI Imaging
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Imaging the Bile Duct With the OFDI Probe
Description: The number of subjects in which the performed OFDI imaging visualizes common bile duct and common hepatic duct strictures.
Time Frame: day 1, during diagnostic procedure
Population: Seven subjects were enrolled and imaged in this study
Measure: Count of Participants; unit: Participants
Groups:
- Optical Frequency Domain Imaging (OFDI Imaging: Subject will swallow an OFDI capsule and images will be obtained using MGH Optical Frequency Domain Imaging (OFDI) imaging system.
  MGH Optical Frequency Domain Imaging (OFDI): Imaging of biliary tract with OFDI system using MGH Optical Frequency Domain Imaging (OFDI) System
Arm/Group | Optical Frequency Domain Imaging (OFDI Imaging
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Arm/Group | OFDI Imaging
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No